CLINICAL TRIAL: NCT06124053
Title: Comparing Outcomes of Group Voice Therapy and Individual Voice Therapy in Children With Dysphonia Between the Ages of 7-11
Brief Title: Investigation of the Effectiveness of Group Voice Therapy in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Özlem Beşik Topçu, Principal Investigator, Hacettepe University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUSLP_GROUPVOICETHERAPY
Record Dates: First submitted 2023-10-16; First posted 2023-11-09 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Dysphonia
Keywords: voice therapy; group voice therapy; pediatric voice disorders; pediatric voice therapy
MeSH Terms: conditions — Dysphonia

STUDY DESIGN:
Intervention Model Description: Participants will be grouped based on the Grade scores on the GRBAS scale using a stratified sampling method.
Who Masked: Outcomes Assessor
Masking Description: The allocation of participants to groups will be carried out through stratified sampling based on the Grade parameter of the GRBAS scoring. Accordingly, individuals conducting GRBAS scoring will listen to the recordings of participants in an anonymous manner.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group Voice Therapy (Experimental): In this research, a total of eight sessions of "group voice therapy" will be applied as the intervention approach. It is planned that each group will consist of three participants. Participants will be evaluated before the intervention, after the intervention, at the third-month follow-up assessment, and at the sixth-month follow-up assessment. Both formal and informal assessment tools have been preferred for the evaluation. Researchers will collect case histories and demographic information. For the acoustic assessment of the participants, voice recordings will be obtained through the ComputerizedSpeech Lab (CLS) program. GRBAS scores will be conducted by the researchers, while Pediatric Voice Handicap Index (pVHI) and Pediatric Voice Related Quality of Life (pVRQOL) scales will be filled out by parents.
  Interventions: Behavioral: Group Voice Therapy
- Individual Voice Therapy (Active Comparator): In this research, a total of eight sessions of "individual voice therapy" will be implemented as the intervention approach. Participants will be evaluated before the intervention, after the intervention, at the third-month follow-up assessment, and at the sixth-month follow-up assessment. Both formal and informal assessment tools have been chosen for the evaluation. Researchers will collect case histories and demographic information. For the acoustic assessment of the participants, voice recordings will be obtained through the CLS program. GRBAS scores will be conducted by the researchers, while pVHI and pVRQOL scales will be filled out by parents or guardians.
  Interventions: Behavioral: Individual Voice Therapy
- Vocal Hygiene Education (Active Comparator): Participants will receive a one-session "vocal hygiene training." Participants will be evaluated twice: once before the vocal hygiene training and again 8 weeks after the vocal hygiene training. Both formal and informal assessment tools have been preferred for the evaluation. Researchers will collect case histories and demographic information. For the acoustic assessment of the participants, voice recordings will be obtained through the CLS program. GRBAS scores will be conducted by the researchers, while pVHI and pVRQOL scales will be filled out by parents.
  Interventions: Behavioral: Vocal Hygiene Education

INTERVENTIONS:
Behavioral: Group Voice Therapy — The "group voice therapy" intervention consists of a total of eight sessions. The session contents include both direct and indirect voice therapy approaches. Each group is composed of three participants. The session durations are planned to be 45-60 minutes each.
  Arms: Group Voice Therapy
Behavioral: Individual Voice Therapy — The "individual voice therapy" intervention consists of a total of eight sessions. The session contents include both direct and indirect voice therapy approaches. The session durations are planned to be 45-60 minutes each.
  Arms: Individual Voice Therapy
Behavioral: Vocal Hygiene Education — Regarding vocal hygiene training, information related to voice production and respiratory characteristics will be provided, and guidance on correct and incorrect voice use will be given.
  Arms: Vocal Hygiene Education

SUMMARY:
This study aims to investigate whether there is a difference between groups receiving "group voice therapy" and "individual voice therapy" in pediatric populations diagnosed with dysphonia. In this context, the goal is to comprehensively examine the effectiveness of "group voice therapy" in pediatric populations compared to similar studies in the literature. In line with this objective, it is aimed to comprehensively test its effectiveness by including perceptual and acoustic evaluation findings, objective and subjective assessments, and incorporating comparison and control groups into the study, as compared to similar studies in the literature.

DETAILED DESCRIPTION:
There are three groups in total in the study: two research groups and one control group. The first research group will receive "group voice therapy". Group voice therapy sessions are arranged in groups of three. A total of eight sessions will be given, one session per week. The second research group will receive "individual voice therapy". In this context, participants will be given individual voice therapy for a total of eight sessions, one session per week. The voice therapy approach to be applied to participants receiving individual voice therapy and group voice therapy includes direct and indirect voice therapy methods.Control group participants will receive a one-session "vocal hygiene training".

Control group participants will be evaluated before and after vocal hygiene training. The first and second research groups will be evaluated four times in total: before therapy, after therapy, third month follow-up and sixth month follow-up. It is aimed to examine the effectiveness of "group voice therapy" by comparing the findings obtained from the approaches. Objective and subjective evaluation tools will be used in the evaluations. It is expected that Research Group 1, receiving "group voice therapy," and Research Group 2, receiving "individual voice therapy," will demonstrate a significant decrease in the primary outcome measure, the GRBAS score, and secondary outcome measures, including the Pediatric Voice Handicap Index score, the Teacher's Perception-Based Voice Handicap Index score, and a significant increase in the Pediatric Voice-Related Quality of Life Scale score when comparing pre-therapy and post-therapy assessments. It is anticipated that these significant changes will be sustained in the follow-up evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with vocal fold lesions.
* Being referred to Hacettepe University Speech and Language Therapy Department for a diagnosis of voice disorder by Hacettepe University Ear, Nose, and Throat Department.
* Being in the age range of 7-11.
* Having Turkish as the native language.

Exclusion Criteria:

* Having a history of any upper respiratory tract infection up to two weeks before the date of data collection (it is requested to consider the last two weeks as a reference in one of the questionnaires to be filled out).
* Having any known neurological, systemic, or endocrinological disease that affects one's voice.
* Having undergone any surgical intervention related to the voice or received voice therapy before the research process.
* Having a diagnosis of current hearing loss.
* Having a neurological or psychiatric diagnosis.
* The family or child not wanting to participate in the study.
* Not having acquired reading and writing skills yet

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes observed in the GRBAS score | Change from the baseline to tenth week
  The changes observed in the GRBAS parameters between pre-intervention and post-intervention evaluations.
Changes observed in the GRBAS score | Change from the baseline to third month follow-up evaluation
  The changes observed in the GRBAS parameters between pre-intervention and post-intervention evaluations.
Changes observed in the GRBAS score | Change from the baseline to sixth month follow-up evaluation
  The changes observed in the GRBAS parameters between pre-intervention and post-intervention evaluations.

SECONDARY OUTCOMES:
The change observed in the Pediatric Voice Handicap Index score | Change from the baseline to tenth week
  The changes observed in the Pediatric Voice Handicap Index total score and subscale scores between pre-intervention and post-intervention evaluations.
The change observed in the Pediatric Voice Related Quality of Life score | Change from the baseline to tenth week
  The changes observed in the Pediatric Voice Quality of Life score and scores between pre-intervention and post-intervention evaluations.
Change in Acoustic Voice Characteristics | Change from the baseline to tenth week
  The changes observed in the F0, Jitter, Shimmer, and Noise to Harmonic Ratio values for the sustain /a/ phonation recording obtained through the Multi-Dimensional Voice Program (MDVP) by Kaypentax Computerized Speech Lab between pre-therapy and post-therapy evaluations.
The change observed in the Pediatric Voice Handicap Index score | Change from the baseline to third month follow-up evaluation
  The changes observed in the Pediatric Voice Handicap Index total score and subscale scores between pre-intervention and post-intervention evaluations.
The change observed in the Pediatric Voice Related Quality of Life score | Change from the baseline to third month follow-up evaluation
  The changes observed in the Pediatric Voice Quality of Life score and scores between pre-intervention and post-intervention evaluations.
Change in Acoustic Voice Characteristics | Change from the baseline to third month follow-up evaluation
  The changes observed in the F0, Jitter, Shimmer, and Noise to Harmonic Ratio values for the sustain /a/ phonation recording obtained through the Multi-Dimensional Voice Program (MDVP) by Kaypentax Computerized Speech Lab between pre-therapy and post-therapy evaluations.
The change observed in the Pediatric Voice Handicap Index score | Change from the baseline to sixth month follow-up evaluation
  The changes observed in the Pediatric Voice Handicap Index total score and subscale scores between pre-intervention and post-intervention evaluations.
The change observed in the Pediatric Voice Related Quality of Life score | Change from the baseline to sixth month follow-up evaluation
  The changes observed in the Pediatric Voice Quality of Life score and scores between pre-intervention and post-intervention evaluations.
Change in Acoustic Voice Characteristics | Change from the baseline to sixth month follow-up evaluation
  The changes observed in the F0, Jitter, Shimmer, and Noise to Harmonic Ratio values for the sustain /a/ phonation recording obtained through the Multi-Dimensional Voice Program (MDVP) by Kaypentax Computerized Speech Lab between pre-therapy and post-therapy evaluations.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma ESEN AYDINLI, Assoc. Prof., Study Chair — Hacettepe University, Speech and Language Therapy Departmant; Meltem Çiğdem KİRAZLI, Ph.D., Study Chair — Hacettepe University, Speech and Language Therapy Departmant; Taner Yılmaz, Prof., Study Chair — Hacettepe University, Department of Otorhinolaryngology
Locations (1):
- Hacettepe University, Speech and Language Therapy, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No